CLINICAL TRIAL: NCT07015918
Title: A PHASE 1, OPEN-LABEL, 2-PERIOD, FIXED-SEQUENCE STUDY TO INVESTIGATE THE ABSORPTION, DISTRIBUTION, METABOLISM, AND EXCRETION OF [14C]PF-07976016 AND TO ASSESS THE ABSOLUTE BIOAVAILABILITY AND FRACTION ABSORBED OF PF-07976016 IN HEALTHY MALE PARTICIPANTS USING A [14C]-MICROTRACER APPROACH
Brief Title: A Study to Understand How the Study Medicine (PF-07976016) is Processed and Eliminated in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C5541002; 2024-518535-11-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Participants will receive doses of PF-07976016 with and without radiolabel.
  Interventions: Drug: [14C] PF-07976016; Drug: PF-07976016

INTERVENTIONS:
Drug: [14C] PF-07976016 — [14C] PF-07976016 liquid (oral) formulation
Drug: PF-07976016 — PF-07976016 liquid (oral) formulation
Drug: [14C] PF-07976016 — [14C] PF-07976016 intravenous (IV) formulation

SUMMARY:
The purpose of this study is to learn about how much the study medicine PF-07976016 will be taken up and processed by healthy male participants. The total number of weeks of the study is up to approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males, 18 to 65 years of age
* BMI 17.5 to 32 kg/m2 and a total body weight >50 kg (110 lb)
* Willing and able to comply with all study procedures

Exclusion Criteria:

* History of irregular bowel movements or lactose intolerance
* Any medical or psychiatric condition or laboratory abnormality or other condition that may increase the risk of study participation
* Use of any prohibited or concomitant medication(s)
* Presence of specified abnormalities on diagnostic assessments including clinical laboratory tests
* Positive urine drug test
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence
* Use of tobacco/nicotine containing products in excess of the equivalent of 5 cigarettes/day
* Previous administration of an investigational product within 30 days preceding the first dose of study medicine in this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male participants
Enrollment: 8 (Actual)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Total recovery of radioactivity expressed as a percent of total oral radioactive dose administered. | From dose (Day 1) and for up to 21 days thereafter

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | First dose (Day 1) through 28 to 35 days after final dose (approximately 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5541002